CLINICAL TRIAL: NCT03828136
Title: Safety and Effectiveness of Novum Vitrium® Cervical Cage in Anterior Cervical Discectomy and Fusion. A Randomized, Controlled, Non-inferiority, Pivotal Study
Brief Title: Novum Vitrium® Cervical Cage in Anterior Cervical Discectomy and Fusion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor business decision
Sponsor: Bio2 Technologies (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT-17-001
Record Dates: First submitted 2019-01-25; First posted 2019-02-04 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Symptomatic Cervical Disc Disease
Keywords: Cervical Disc Disease; ACDF; Single-level
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: A total of 168 patients will be randomized in 7:2 ratio to Investigational (n=130) and Control arms (n=38).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ACDF with Novum Vitrium® Cervical Interbody Device (Experimental): A resorbable cervical interbody cage.
  Interventions: Device: Novum Vitrium® Cervical Interbody Device
- ACDF with Allograft (Active Comparator): Structural allograft made from structural corticocancellous allograft bone.
  Interventions: Device: Allograft Ring or Block

INTERVENTIONS:
Device: Novum Vitrium® Cervical Interbody Device — For spinal fusion procedure at one level (C3 to T1) of the cervical spine.
  Other Names: Novum Vitrium® Cervical Cage
  Arms: ACDF with Novum Vitrium® Cervical Interbody Device
Device: Allograft Ring or Block — Standard of Care
  Arms: ACDF with Allograft

SUMMARY:
A prospective, multicenter, randomized, concurrently controlled, noninferiority clinical trial to compare the safety and effectiveness of instrumented Bio2 Vitrium Cervical Interbody Device in anterior cervical discectomy and fusion (ACDF) with structural allograft bone and local autologous bone graft in treating patients with a symptomatic degenerative cervical disc disease at one level from C3/C4 to C7/T1.

DETAILED DESCRIPTION:
The study will evaluate if Bio2 Vitrium® Cervical Interbody Device (VCIBD) is non-inferior to allograft cage in single-level ACDF with the use of local autologous bone. VCIBD is a restorable cervical interbody cage for the treatment of fusion, following discectomy, of the cervical spine from C3/C4 disc space to the C7/T1 disc space. The material used to manufacture the implant is 13-93 bioactive glass, which is a silicate-based material as described in ASTM F1538-03(R2017). The implant has high porosity and strength and does not contain any biological material or constitute a combination product. The device has a central lumen for packing with autograft. VCIBD is intended to be used with a supplemental fixation system.

The device, when placed between the vertebrae, provides mechanical stability and prevents subsidence prior to bone ingrowth. It restores and maintains the intervertebral space during the fusion process. The porosity and material characteristics provide an osteoconductive matrix that supports bone ingrowth. Additional stabilization is provided by supplemental fixation using anterior cervical plate. The implant incorporates a central lumen, which allows for the cage to be packed with autogenous bone graft.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic cervical disc disease (SCDD) in the one vertebral level between C3/C4 to C7/T1, defined as neck or arm (radicular) pain, or functional or neurological deficit and correlated with radiculopathy or myelopathy or radiographic confirmation (by CT, MRI, x-ray, etc.) of any of the following:

   * Herniated nucleus pulposus;
   * Spondylosis (defined by the presence of osteophytes); or
   * Loss of disc height.
2. Requires only one cervical vertebral level to be surgically treated, confirmed radiologically by Xray, CT, or MRI and correlated with neurologic examination prior to enrollment;
3. Age between 22 and 70 years (inclusive);
4. Skeletally mature patients;
5. Failed at least 6 weeks of conservative treatment (e.g. medication, physical therapy), or exhibit progressive symptoms or signs of spinal cord/nerve root compression with continued non-operative care;
6. Neck Disability Index (NDI) Questionnaire score of at least 30 (on a scale from 0 to 100);
7. Able to read and Understand all documents used in this study, including the Informed Consent and patient-reported outcome questionnaires;
8. Understand and read English at elementary level;
9. Patient must understand and sign the Informed Consent document that has been approved by the Ethics committee, Institutional review Board and the FDA.

Exclusion Criteria:

1. More than one vertebral level requiring treatment, confirmed radiologically by X-ray, CT, or MRI
2. Cervical instability;
3. Prior fusion surgery at any cervical vertebral level;
4. Prior surgery at the level to be treated with the exception of surgery that does not require the use of hardware and/or the treatment of facet disease;
5. Severe facet disease;
6. Clinically compromised vertebral bodies at the affected level(s) due to current or past trauma
7. Neck or arm pain of unknown etiology;
8. Osteoporosis, osteopenia, Paget's disease, osteomalacia or any other metabolic bone disease;

   a. Osteoporosis is defined as history of fragility fracture and Dexa (DXA) T-score < -2.5 or QCT T-score < 80mg/cubic cm. History of a fragility fracture requires that a DXA scan or QCT scan is completed
9. Pregnant or interested in becoming pregnant in the next 2 years;
10. Active systemic or local infection;
11. History of severe allergy or anaphylaxis especially to titanium, polyethylene, cobalt, chromium or molybdenum;
12. Taking medications or any drug known to potentially interfere with bone/soft tissue healing (e.g., steroids, bisphosphonates);
13. Rheumatoid arthritis or another autoimmune disease that affects musculoskeletal system;
14. Acquired immune deficiency syndrome (AIDS) or an AIDS-related complex;
15. Active malignancy or history of invasive malignancy within the last five years, except for superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitely treated; patients with carcinoma in situ of the uterine cervix treated definitely more than 1 year prior to enrollment may enter the study;
16. Neuromuscular disorders such as muscular dystrophy, spinal muscular atrophy, and amyotrophic lateral sclerosis;
17. Pre-existent neurologic or mental disorder which would preclude accurate evaluation and followup (i.e. Alzheimer's disease, Parkinson's disease, unstable psychiatric disorder with hallucinations and/or delusions or schizophrenia);
18. Substance use disorder categorized as moderate to severe as defined in DSM-V;
19. Mental/Psychiatric disorder as defined in DSM-V;
20. Alcohol abuse disorder categorized as moderate to severe as defined in DSM-V;
21. Current Smokers;
22. Use of bone growth stimulator in the region of the cervical spine within the past 30 days;
23. Participation in other investigational device or drug clinical trials within 30 days of surgery;
24. Prisoners;
25. Morbid obesity, defined as body mass index ("BMI") > 40;
26. Type 1 diabetes mellitus requiring daily insulin therapy unless there is documentation of a recent A1c (within 6 months) of less than 7.1 or Type 2 diabetes where the clinical presentation precludes the patient from having surgery;
27. Involved in litigation related to the spine;
28. On workers compensation

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Number of participants who have achieved of radiologic fusion assessed by roentgenographic examination. | 12 months
  Successful fusion is based on meeting the roentgenographic examination criteria showing the evidence of: bridging trabecular bone between the involved motion segments; translation motion <3mm; and angular motion ≤2°.
Change in Neck Disability Index (NDI) with a response greater than or equal to 15 from baseline. | 12 months
  NDI consists of ten items addressing function activities, pain intensity, concentration, and headache.It has a continuous various with a range from 0 (best) to 100 (worse). The effectiveness endpoint is the difference between the baseline value and the follow-up (12 month) value.
Number of participants with neurological success. | 12 months
  Neurological success is a binary outcome as follows:
  * Maintenance or improvement of the neurological status;
  * Worsening of the neurological status.
  Worsening of the neurological status is defined as permanent new neurologic damage or permanent new nerve root injury related to the surgically treated level, defined as one or more:
  * Permanent decrease in one or more grades of motor strength compared to baseline;
  * Permanent new sensory deficit (paresthesia or anesthesia) in a specific cervical nerve root distribution.
Number of participants who have completed follow-up up to month 12 without Secondary Surgical Intervention (SSI). | 12 months
  Identified as the absence of revision, removal, reoperation, or supplemental fixation at the index level

SECONDARY OUTCOMES:
Measurement of Pain at neck and at arm and shoulder as assessed by Visual Analog Scale | 6, 12, and 24 months
  Neck pain and arm/shoulder pain as measured by the Visual Analog Scale (VAS) on the scale from 0 (no pain) to 100 (worst imaginable pain)
Quality of Life assessed by 36-Item Short Form Health Survey Version 2 (SF-36v2) | 6, 12, and 24 months
  The SF-36v2 Health Survey is a 36-item instrument for measuring health status and outcomes. It yields an eight-scale profile score from the following eight health concepts: physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and general mental health (psychological distress and psychological well being). In addition, two composites scores are constructed using factorial modeling, one from physical health composite score (PCS) and one for mental health composite score (MCS).
Quality of Life assessed by EuroQoL Health Related Quality of Life - 5 Dimensions - 3 Levels (EQ-5D-3L) | 6, 12, and 24 months
  The EQ-5D-3L is a standardized instrument used as a measure of health outcomes. It contains questions in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and provides a simple descriptive profile and single index for health status preference. In addition, there is a Visual Analog Scale (VAS). The VAS is the participant's rating of their health on a scale of 0 "worst imaginable health state" to 100 "best imaginable health state".
Measurement of the use of Pain Medication for Cervical Spine. | 6, 12, and 24 months
  The use of prescription and OTC pain medication for cervical spine-related pain will be recorded in addition to the use of opioids on study-specific logs.
Measurement of Patient Satisfaction: patients to rate their satisfaction | 6, 12, and 24 months
  Developed based on IDE spine studies. It asks patients to rate their satisfaction with their treatment (6 choices from "Very Satisfied" to "Very Dissatisfied"), and question regarding every day activities and their ability to complete them. There are 5 choices from "Definitely" to "Definitely Not".

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Orthopaedic Education and Research Institute, Orange, California
  - Hartford Hospital, Hartford, Connecticut
  - Indiana Spine Group, Carmel, Indiana
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - Upstate Medical University, Syracuse, New York
  - M3-Emerging Medical Research, Durham, North Carolina
  - Arise Medical Center, Austin, Texas